CLINICAL TRIAL: NCT00459381
Title: A Phase II Trial of GW786034 (Pazopanib) in Patients With Recurrent Glioblastoma
Brief Title: Pazopanib in Treating Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02710; NABTC-0602; U01CA062399 (NIH); CDR0000538083 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive oral pazopanib hydrochloride daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Other: laboratory biomarker analysis
  Interventions: Drug: pazopanib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given orally
  Other Names: GW786034B; Votrient
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well pazopanib works in treating patients with recurrent glioblastoma. Pazopanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the therapeutic efficacy of pazopanib hydrochloride, as measured by 6-month progression-free survival (PFS), in patients with recurrent glioblastoma.

II. Determine the safety profile of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the efficacy of this drug, as measured by radiographic response, time to progression, and overall survival, in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral pazopanib hydrochloride daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme, including gliosarcoma

  * Recurrent disease
* Must have unequivocal radiographic evidence of tumor progression by MRI, as defined by any of the following:

  * 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline
  * Clear worsening of any evaluable disease
  * Appearance of any new lesions or site
  * Clear clinical worsening
* Must have failed prior radiotherapy that was completed ≥ 42 days ago
* Patients who received prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease, rather than radiation necrosis, based on positron emission tomography (PET) scan, thallium scanning, magnetic resonance spectroscopy, or surgical documentation of disease
* Treatment for no more than 2 prior relapses allowed

  * Relapse is defined as progression following initial therapy (i.e., radiotherapy with or without chemotherapy, if that was used as initial therapy; therefore no more than 3 prior therapies [initial therapy and therapy for 2 relapses] allowed)

    * If the patient had a surgical resection for relapsed disease and no anticancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse
    * For patients who had prior therapy for a low-grade glioma, the surgical diagnosis of a glioblastoma multiforme will be considered the first relapse
* Karnofsky performance status 60-100%
* Life expectancy > 8 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 10 g/dL (may be reached by transfusion)
* Platelet count ≥ 100,000/mm^3
* PT/INR/PTT ≤ 1.2 times upper limit of normal (ULN)
* SGOT < 2.5 times ULN
* Bilirubin < 2.5 times ULN
* Creatinine < 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Urine protein:creatinine ratio > 1 OR urine protein < 1,000 mg by 24-hour urine collection OR proteinuria < 1+
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during study therapy OR practice abstinence from sexual intercourse for 14 days prior to, during, and for ≥ 21 days after study therapy
* Systolic blood pressure (BP) ≤ 140 mm Hg and diastolic BP ≤ 90 mm Hg

  * Prior initiation or adjustment of BP medication allowed provided the average of 3 BP readings is ≤ 140/90 mm Hg
* No uncontrolled significant medical illnesses that would preclude study therapy
* No other conditions, including any of the following:

  * Serious or nonhealing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * Cerebrovascular accident (CVA) within the past 6 months
  * Myocardial infarction, cardiac arrhythmia, admission for unstable angina, cardiac angioplasty, or stenting within the past 84 days
  * Venous thrombosis within the past 84 days
  * New York Heart Association (NYHA) class III or IV heart failure

    * Asymptomatic NYHA class II heart failure while on treatment allowed
* No other cancer except for nonmelanoma skin cancer or carcinoma in situ of the cervix unless in complete remission and off of all therapy for that disease for ≥ 3 years
* No disease that would obscure toxicity or dangerously alter drug metabolism
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to pazopanib hydrochloride or other agents
* No QTc prolongation (i.e., QTc interval ≥ 500 msecs) or other significant ECG abnormalities
* No condition that impairs the ability to swallow and retain pazopanib hydrochloride, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* See Disease Characteristics
* Recovered from prior therapy
* At least 28 days since prior resection of recurrent or progressive tumor and recovered

  * Residual disease after resection of recurrent glioblastoma is not mandated for eligibility into the study
* More than 7 days since prior noncytotoxic agents (e.g., interferon, tamoxifen, thalidomide, or isotretinoin)

  * Radiosensitizers allowed
* More than 14 days since prior investigational agents
* More than 14 days since prior vincristine
* More than 21 days since prior procarbazine
* More than 28 days since prior cytotoxic therapy
* More than 42 days since prior nitrosoureas
* No prior bevacizumab
* No prior sorafenib tosylate or sunitinib malate
* No prior pazopanib hydrochloride
* No concurrent CYP2C9 substrates, including any of the following:

  * Anticoagulants (e.g., warfarin [therapeutic doses only])
  * Oral hypoglycemics (e.g., glipizide, glyburide, tolbutamide, glimepiride, or nateglinide)
  * Ergot derivatives (e.g., dihydroergotamine, ergonovine, ergotamine, or methylergonovine)
  * Neuroleptics (e.g., pimozide)
  * Erectile dysfunction agents (e.g., sildenafil, tadalafil, or vardenafil)
  * Antiarrhythmics (e.g., bepridil, flecainide, lidocaine, mexilitine, amiodarone, quinidine, or propafenone)
  * Immune modulators (e.g., cyclosporine, tacrolimus, or sirolimus)
  * Miscellaneous drugs (e.g., theophylline, quetiapine, risperidone, tacrine, clozapine, or atomoxetine)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy (including chemotherapy, radiotherapy, hormonal treatment, or immunotherapy) or investigational drugs
* No concurrent enzyme-inducing anti-epileptic drugs (EIAEDs)

  * Non-EIAEDs allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fine, MD, Principal Investigator — North American Brain Tumor Consortium
Locations (9):
- United States (9):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - National Cancer Institute Neuro-Oncology Branch, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwamoto FM, Lamborn KR, Robins HI, Mehta MP, Chang SM, Butowski NA, Deangelis LM, Abrey LE, Zhang WT, Prados MD, Fine HA. Phase II trial of pazopanib (GW786034), an oral multi-targeted angiogenesis inhibitor, for adults with recurrent glioblastoma (North American Brain Tumor Consortium Study 06-02). Neuro Oncol. 2010 Aug;12(8):855-61. doi: 10.1093/neuonc/noq025. Epub 2010 Mar 3. PMID 20200024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects accrued between June 2007 to January 2008 at 4 NABTC Cancer Centers using their outpatient facilities. Survival follow-up extended to June 2009
Groups:
- Treatment (Pazopanib Hydrochloride): Patients receive oral pazopanib hydrochloride daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Other: laboratory biomarker analysis
  pazopanib hydrochloride: Given orally
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Pazopanib Hydrochloride)
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 53 [29 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22
Karnofsky Performance Status Scale [Number; unit: participants] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  participants
    90-100 | 26
    60-80 | 9
Prior Radiotherapy [Number; unit: participants] | 35
Time from Radiotherapy to study enrollment [Median (Full Range); unit: months] | 10 [1 to 169]
Number of Prior chemotherapy reginmens [Number; unit: participants]
  1 | 24
  2 | 9
  3 | 2
Surgery for recurrence for current progression prior to enrollment [Number; unit: participants]
  Yes | 8
  No | 27

OUTCOME MEASURES:

1. Primary Outcome: 6 Months Progression-free Survival
Description: Calculated from study registration till 6month time point. Progression defined by Macdonald criteria Progression imaging features: 25% of more increase in enhancing lesions; any new lesions clinical features: clinical deterioration
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
percent | 3 [0.001 to 15]

2. Primary Outcome: Number of Participants Discontinuing Treatment Due to Toxicity
Description: Use NCI Common toxicity Criteria Adverse Event Version 3.0 to grade toxicities. Any patient who received at least one dose of pazopanib was evaluable for toxicity. Calculated the number of participants who had an event that was related to pazopanib that caused the patient to stop treatment due to this event.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
Participants
  thrombotic/embolic | 3
  CNS hemorrhage | 1

3. Secondary Outcome: Most Common Toxicities Experienced After at Least One Dose of Pazopanib
Description: NCI Common Toxicity Criteria (CTCAE) version 3.0. All patients that received at least one dose of pazopanib were evaluable. All events recorded that were related to drug were calculated per patient.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
percentage of participants
  hypertension | 37
  fatigue | 34
  elevated ALT | 40

4. Secondary Outcome: Overall Radiographic Response (ORR) Rate
Description: The Macdonald criteria, roughly similarly to other systems, divides response into 4 types of response based on imaging (MRI) and clinical features
  1: complete response; 2: partial response; 3:stable disease; 4:progression
  Complete response imaging features: disappearance of all enhancing disease (measurable and non-measurable) sustained for at least 4 weeks; no new lesions clinical features; no corticosteroids; clinically stable or improved
  Partial response imaging features: 50% or more decrease of all measurable enhancing lesions sustained for at least 4 weeks: no new lesions clinical features: stable or reduced corticosteroids; clinically stable or improved
  Stable disease imaging features: does not qualify for complete response, partial response or progression clinical features: clinically stable
  Progression imaging features: 25% of more increase in enhancing lesions; any new lesions clinical features: clinical deterioration
Time Frame: 2 years
Population: 34 pts had follow-up scans and wee evaluable for objective radiographic response (ORR)
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 34
percent | 5.9 [0.7 to 21]

5. Secondary Outcome: Best Radiographic Response
Description: Using the Macdonald criteria, the best MRI image response while the patient was on active treatment.
  1: complete response; 2: partial response; 3:stable disease; 4:progression
  Complete response imaging features: disappearance of all enhancing disease (measurable and non-measurable) sustained for at least 4 weeks; no new lesions clinical features; no corticosteroids; clinically stable or improved
  Partial response imaging features: 50% or more decrease of all measurable enhancing lesions sustained for at least 4 weeks: no new lesions clinical features: stable or reduced corticosteroids; clinically stable or improved
  Stable disease imaging features: does not qualify for complete response, partial response or progression clinical features: clinically stable
  Progression imaging features: 25% of more increase in enhancing lesions; any new lesions clinical features: clinical deterioration
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 34
percentage of participants
  Progressive Disease | 32
  Stable Disease | 62
  Partial Response | 6

6. Secondary Outcome: Overall Survival
Description: calculated from study registration until date of death or patient censored at the last date known alive
Time Frame: From date of registration to date of death due to any cause, assessed up to 2 years
Population: All 35 patients were included in an intent to treat analysis for PFS and OS.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
weeks | 35 [24 to 47]

7. Secondary Outcome: Time to Progression or Progression Free Survival
Description: PFS for patients who died on treatment or within 30 days of the end of treatment w/out progression date, was date of death. All other pts without documented progression were censored at the date of last follow-up prior to start new treatment.
  All 35 patients were included in an intent to treat analysis for PFS and OS. 3 pts censored for PFS, all less than 2 wks after study registration.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
weeks | 12 [8 to 14]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (Pazopanib Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 35/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride) (N=35)
anemia (Blood and lymphatic system disorders) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 7 (7)
lymphopenia (Blood and lymphatic system disorders) | 12 (12)
neutropenia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Investigations) | 9 (9)
arterial hypertension (Vascular disorders) | 13 (13)
fatigue (General disorders) | 12 (12)
weight loss (Investigations) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 5 (5)
abdominal distension (Gastrointestinal disorders) | 2 (2)
flatulence (Gastrointestinal disorders) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 4 (4) — heartburn
Intracranial hemorrhage (Nervous system disorders) | 3 (3)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
elevated ALT (Investigations) | 14 (14)
elevated AST (Investigations) | 8 (8)
hyperbilirubinemia (Investigations) | 7 (7)
hypermagnesemia (Metabolism and nutrition disorders) | 3 (3)
hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
proteinuria (Metabolism and nutrition disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 2 (2)
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less